CLINICAL TRIAL: NCT05005169
Title: Cost-consequence Analysis of Intrapartum Streptococcal B Detection by PCR Versus Antenatal Culture at 35-38 SA in the Optimization of Intrapartum Antibiotic Prophylaxis
Brief Title: CCA of SGB PCR Versus SGB Culture at 35-38 SA in the Optimization of Intrapartum Antibiotic Prophylaxis
Acronym: DEPIST2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: RC20_0069
Record Dates: First submitted 2021-05-20; First posted 2021-08-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Streptococcus Agalactiae
Keywords: Health economics, streptococcus B, screening, PCR
MeSH Terms: conditions — Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrapartum streptococcal B detection by PCR (Experimental): The automatons will be installed by the laboratory in the delivery rooms and used delocalized by the obstetrical teams. Verification and validation of results will be ensured by the microbiology laboratory team, according to the recommendations and procedures already in use for off-site biology.
  Interventions: Diagnostic Test: SGB PCR
- intrapartum streptococcal B detection by "SGB culture" strategy (Active Comparator)
  Interventions: Diagnostic Test: SGB culture

INTERVENTIONS:
Diagnostic Test: SGB PCR — This is a multi-center, randomized cluster and crossover study, and is open-label. The cluster is defined by the hospital center. Each center will therefore experiment with both strategies and the hospital centers will be randomized according to two arms:
  * Arm n°1 : 1st period with "SGB culture" strategy and 2nd period with "SGB PCR" strategy.
  * Arm n°2 : 1st period with "SGB PCR" Strategy and 2nd period with "SGB culture" Strategy Each inclusion period will last 6 weeks, with a 1-month wash-in period before each of the two inclusion periods of the study (training of the teams in intrapartum PCR detection). A wash-out period is not necessary in this study because the PCR machine will be removed from the centers when switching to the GBS culture strategy.
  During these two periods, all patients meeting the inclusion and non-inclusion criteria will be included in the study after presentation of the study and oral consent.
  Other Names: Test Xpert® SGB and GeneXpert® Systems / GeneXpert® IV System (GX-4) - CEPHEID
  Arms: intrapartum streptococcal B detection by PCR
Diagnostic Test: SGB culture — This is a multi-center, randomized cluster and crossover study, and is open-label. The cluster is defined by the hospital center. Each center will therefore experiment with both strategies and the hospital centers will be randomized according to two arms:
  * Arm n°1 : 1st period with "SGB culture" strategy and 2nd period with "SGB PCR" strategy.
  * Arm n°2 : 1st period with "SGB PCR" Strategy and 2nd period with "SGB culture" Strategy Each inclusion period will last 6 weeks, with a 1-month wash-in period before each of the two inclusion periods of the study (training of the teams in intrapartum PCR detection). A wash-out period is not necessary in this study because the PCR machine will be removed from the centers when switching to the GBS culture strategy.
  During these two periods, all patients meeting the inclusion and non-inclusion criteria will be included in the study after presentation of the study and oral consent.
  Arms: intrapartum streptococcal B detection by "SGB culture" strategy

SUMMARY:
Early-onset neonatal infection (EONI), occur within 7 days of birth. They are most often due to Streptococcus B (GBS) and are associated with heavy and costly morbidity and mortality. The strategy combining antenatal detection (PV9) of GBS colonization and intrapartum antibiotic therapy has led to a spectacular decrease in the number of GBS EONI's that have become rare (0.3/1000 births). Current detection is based on the culture of a vaginal swab taken between 35 and 38 SA. Because the positive predictive value of PV9 compared to a culture on the day of delivery is 60%, two problems persist: i) 20% of women and newborns are sometimes unnecessarily exposed to antibiotics with known short-term and long-term harmful effects; ii) more than half of newborns developing EONI are born to mothers with negative PV9. There is a risk of not treating intrapartum colonization when PV9 is negative, and overtreating an uncolonized PV9-positive woman at the time of delivery. These inappropriate antibiotic therapies generate additional maternal-fetal care, examinations, treatments and hospitalizations with significant costs.

Today, a feasible, rapid, sensitive (90-95%) and specific (95-98%) PCR test (Xpert GBS, CEPHEID) can be used to detect women colonized with GBS at the beginning of labor. A recent study (submitted for publication) including 782 women with risk factors for infection (intrapartum fever or prolonged rupture of membranes) who were subjected to PV9 and intrapartum PCR (IP PCR), identified 19% potential reclassification of GBS status, with a potential saving of 6% intrapartum antibiotic.

We postulate that the replacement of PV9 by the generalized use of GBS intrapartum detection would optimize the indications for intrapartum antiobiotherapy, avoiding (i) unnecessary and deleterious care consumption in the absence of intrapartum GBS colonization, and (ii) avoidable EONIs occurring in the absence of intrapartum antiobiotherapy when GBS colonization has not been diagnosed.

We propose to conduct a cost-consequence study because the criteria for clinically relevant judgments do not allow for cost-effectiveness or cost-utility analysis. Indeed, the intrapartum PCR strategy has consequences for both mother and child and these consequences cannot be aggregated.

Thus, cost-consequence analysis based on criteria validated by clinicians and the literature seemed to us to be the most pragmatic approach and the most likely to help public decision making.

The objective of this work is therefore to carry out a cost-consequence analysis comparing the intrapartum antibiotic prophylaxis strategy based on intrapartum GBS colonization screening by PCR, with the current strategy based on antenatal screening by culture between 35 and 38 SA.

DETAILED DESCRIPTION:
• Inclusion visit : The patient is included in the "GBS culture" group or in the "GBS PCR" group determined by the randomization of the hospital in which she gives birth.

A sample to perform the GBS PCR will be taken or not depending on the strategy in place in the center at the time of inclusion. The patient's management will be adapted according to the test result. The administration of intrapartum antibiotic therapy will be decided by the clinician in charge of the patient based on the result of antenatal GBS screening (PCR or culture) and taking into account the risk factors for EONI. In the GBS PCR group, the clinician will not have access to the result of the antenatal detection, even if the result is forgotten or technically impossible.

• M1 follow-up visit (+/-5 days) by phone The study coordinator will follow up the patient by phone.

The data collected are as below:

* Neonatal infection occurring within the first 6 days of life (this diagnosis requires hospital treatment by intravenous route, and will be verified on the hospitalization report),
* Endometritis in the first month after birth,
* Maternal and/or newborn antibiotic therapy (which one? how long? in which indication?)
* Hospitalization of the mother and/or newborn (which hospital, which department, how long? for what reason).
* Hospitalization report.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the delivery room from 35SA upwards
* Planned vaginal delivery
* Patients who agreed to participate in the study and gave oral consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Complete dilatation (imminent delivery)
* Scheduled caesarean
* Term < 35 SA
* Death in utero
* Medical termination of pregnancy
* Does not speak French
* Opposition to participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women of childbearing age
Enrollment: 3321 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Comparison of total cost of antenatal culture versus intrapartum PCR screening strategy | Day 30
  Cost-consequence analysis:
  - Comparison of the total cost (collective perspective) of the screening strategy (expressed in euros) by antenatal culture versus intrapartum PCR from PV to 30 days postpartum.

SECONDARY OUTCOMES:
Neonatal morbidity-mortality criterion for NPI composite combining over the first 6 days of life | Day 6
  Neonatal morby-mortality criterion: composite criteria (expressed in %)
Criteria for maternal-fetal exposure to antibiotics | Day 30
  Criteria for materno-foetal exposure to ATB (expressed in %)
Maternal morbidity and mortality criteria at 30 days after delivery | Day 30
  a. Maternal mortality
Proportion of appropriate intrapartum TBAs in the CRP arm compared to what would have been indicated using current recommendations | Day 0
  Intrapartum antibiotic therapy will be considered appropriate if i) PCR+ at time of delivery with intrapartum TBA ii) indeterminate PCRwith 2 risk factors for infection with intrapartum TBA, iii) PCR negative without intrapartum TBA iv) PCR negative or indeterminate with 0 or 1 risk factor for infection without intrapartum TBA. The comparison will focus on the proportion of TBAs administered in the "SGB culture" arm, which will be the state of practice and the reference in this pragmatic study.
Feasibility criteria for the intrapartum GBS PCR screening strategy | Day 0
  1. Feasibility of off-site PCR in the birth room: % of PCRs performed for the entire eligible population
  2. Proportion of complete TBA ≥ 4h before delivery
  3. Frequency of PCR "errors" or "invalids
Net financial benefit (cost difference, annually and over 5 years) between different scenarios of dissemination of the strategy considered as efficient (Budget impact analysis; calculation on Excel) | 5 years
  Budget impact analysis allowing to evaluate the net financial benefit of the diffusion of the intrapartum antibiotic prophylaxis strategy based on the screening of GBS colonization in intrapartum by PCR, by comparing scenarios with different rates of development of this strategy, from the National Health Insurance perspective, annually and globally over a 5-year period. This analysis is performed in an Excel sheet, with the following parameters: mean cost of care for this strategy, initial market share of this strategy, expected speed of evolution of its market share compared to other existing strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Christèle Gras-Le Guen, Pr, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - Multon, Nantes, Saint Herblain
  - Gillard, Angers
  - Sentilhes, Bordeaux
  - Houllier, Le Kremlin-Bicêtre
  - Roumieu, Lyon
  - Morel, Nancy
  - Kayem, Paris
  - Anselem, Paris
  - Schmitz, Paris
  - Lassel, Rennes
  - Lecointre, Strasbourg

IPD SHARING:
Plan to Share IPD: No